CLINICAL TRIAL: NCT03673982
Title: Bridging Transitions From Hospital to Home: Collaborative Skill Sharing Intervention With Carers (iCASK)
Brief Title: Carer Skills Training for Inpatients With Anorexia Nervosa (iCASK)
Acronym: iCASK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James Adamson (Other)
Responsible Party: Sponsor-Investigator, James Adamson, Clinical Researcher, South London and Maudsley NHS Foundation Trust
Organization: South London and Maudsley NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPMS ID 33235
Record Dates: First submitted 2017-03-16; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCASK Group (Experimental): Materials and support to aid transitions.
  Interventions: Behavioral: iCASK

INTERVENTIONS:
Behavioral: iCASK — Materials and support to aid transitions

SUMMARY:
To improve treatment for patients with severe anorexia nervosa admitted for inpatient care, and to help their families. Inpatients and their families will be offered a novel intervention which includes multimedia training materials. These materials provide guidance in how families can provide support to maintain and build on changes made during inpatient care

DETAILED DESCRIPTION:
Problem to be solved: Hospital Episode Statistics reveal that admissions for anorexia nervosa are increasing [1]. Admission restores nutrition in a timely manner [2], but psychosocial problems remain and relapse following discharge is common [3]. The mortality post discharge is high [4]. We have found that relapse and bed use post discharge are reduced by a parenting intervention giving the family skills to manage eating disorder behaviours [5].

Innovation: Through a process of co-production, in collaboration with service users and their families, we have developed tools exemplifying emotional coaching behaviour change strategies for patients and their carers (texts, DVDs and podcasts; iCASK programme). These aim of these tools is to improve the transition to outpatient care. These are hosted on a user-friendly, confidential and NHS-compliant platform.

ELIGIBILITY:
Inclusion Criteria:

* aged 17 or over
* DSM-5 diagnosis of Anorexia Nervosa with a body mass index (BMI) of < 18.5 kg/m2

Exclusion Criteria:

* Insufficient knowledge of English
* Severe mental or physical illness needing treatment in its own right (e.g. psychosis or diabetes mellitus)

Ages: 17 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
weight change | at time of admission, at time of discharge (average 12-14 weeks)
  weight change over the admission (weight and height will be combined to report BMI in kg/m^2)

SECONDARY OUTCOMES:
Self-Report Questionnaires to assess psychopathological change for patients over admission and post-discharge. | Questionnaires are administered at time of admission, at time of discharge (average 12-14 weeks) and 3 months post-discharge.
  Battery of quantitative self report measures for patients administered at admission, discharge and 3-month follow up.
  Primary Questionnaire:
  EDEQ (Eating Disorders Questionnaire) - Global score calculated for each time point to assess psychopathological change over time. Reduction in global score would indicate an improvement.
  Secondary Measure: A reduction in scores would indicate an improvement, except for AQ-10 which should remain constant if true Autism detected. Scores will be assessed individually using total scores but then combined with EDEQ to look overall at psychopathological change over time.
  WSAS (Social Adjustment) - Total Score AQ-10 (Autism Quotient) - Total Score indicates levels of autism symptoms. HADS (Anxiety and Depression Scale) - Total Score MR (Motivational Ruler) - Total Score
Self-Report Questionnaires for carers, to assess change in perceived burden over admission and post-discharge. | Questionnaires are administered at time of admission, at time of discharge (average 12-14 weeks) and 3 months post-discharge.
  Battery of quantitative self report measures for carers administered at admission, discharge and 3-month follow up.
  Questionnaire total scores are calculated to provide overview of carer burden. Sub-scales are not used.
  Carer Questionnaires: A decrease in overall scores would indicate an improvement.
  Burden:
  DASS (Depression, Anxiety and Stress Scale) - Total Score used EDSIS (Eating Disorder Symptom Impact Scale) - Total Score used PvAN (Parent vs Anorexia Scale) - Total Score used AESED (accommodation and enabling scale for eating disorders) - Total Score used
Self-Report Questionnaires for carers, to assess change in perceived confidence over admission and post-discharge. | Questionnaires are administered at time of admission, at time of discharge (average 12-14 weeks) and 3 months post-discharge.
  Single quantitative self report questionnaire for carers administered at admission, discharge and 3-month follow up.
  Questionnaire total scores are calculated to provide overview of carer confidence. Sub-scales are not used.
  Carer Questionnaire:
  CASK (Carer Confidence scale) - Total Score used - An increase in score will indicate increased confidence.
Patient satisfaction | at 3 months post-discharge.
  Qualitative feedback from patients, carers and staff - semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Treasure, Prof, Principal Investigator — Principal Investigator
Locations (1):
- Tyson West 2, Bethlem Royal Hospital, Beckenham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No